CLINICAL TRIAL: NCT05690724
Title: A Randomised, Double-blind, Placebo-controlled, Parallel-group Study in Otherwise Healthy Adults With Mild Cognitive Impairment (MCI) Assessing a 16-week Intervention With Mitocholine™, a Functional Food Ingredient
Brief Title: Healthy Adults With Mild Cognitive Impairment (MCI) and a 16-week Intervention With Mitocholine™, a Functional Food Ingredient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mitocholine Ltd (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AFCRO-155
Record Dates: First submitted 2023-01-06; First posted 2023-01-19 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomised, double-blinded, placebo-controlled, parallel proof of concept study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mitocholine™ (Experimental): Mitocholine™ is a novel formulation of three nutrients choline, succinic acid, and nicotinamide (a vitamin B3)
  Interventions: Dietary Supplement: Mitocholine™ or Placebo
- Placebo (Placebo Comparator): The Placebo product will be identical in appearance and taste to the investigational product
  Interventions: Dietary Supplement: Mitocholine™ or Placebo

INTERVENTIONS:
Dietary Supplement: Mitocholine™ or Placebo — Participants will be instructed to consume one bottle of study product daily for the duration of the trial (16 weeks). They will be instructed to consume the product in the morning with breakfast.

SUMMARY:
To evaluate the effect of 16-weeks consumption of Mitocholine on Executive Function and Homocysteine levels in a population experiencing Mild Cognitive Impairment. The study will also include measures of memory, language, S-adenosylmethionone (SAM), Betaine, Choline.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate in the study and comply with its procedures.
2. Able to give written informed consent.
3. Adults aged 55 to 79 years, inclusive.
4. Meet MCI criteria, based on the Peterson criteria (Peterson et al., 1999):

   1. Objective evidence of cognitive impairment as assessed by MoCA (score ≥18 to ≤25).
   2. Absence of major depression as assessed by PHQ (score <10).
   3. Activities of daily living score

      * males ≥4
      * females ≥7
5. Have a homocysteine level ≥11.0μmol/L (Smith D et al, 2018).

Exclusion Criteria:

1. Diagnosis of a major cognitive disorder (e.g. Alzheimer's or Parkinson's disease diagnoses; additionally, confirmation of a mini stroke (TIA) within the last 3 months would be an exclusionary condition).
2. Participants who are pregnant or wish to become pregnant during the trial.
3. Participants who are lactating and/or currently breastfeeding.
4. Participants currently of childbearing potential, but not using an effective method of contraception, as determined by the investigator.
5. Participants with active or a history of alcohol or substance abuse; (exclude elevated Gamma GT & clinically abnormal liver function test).
6. Uncontrolled diabetes (or glycated haemoglobin >7% / 53 mmol/mol).
7. Clinically significant heart, liver, or renal disease (at the discretion of the investigator).
8. Have uncontrolled hypertension SBP > 160mmHg, DBP > 100mmHg).
9. Participants prescribed medications likely to influence memory or mood, as determined by the investigator.
10. Participants with a history of depression (within past 24 months) or any concurrent medical, cognitive or psychiatric condition that would either: compromise his/her ability to comply with the study requirements, may pose significant risk to the participant, or be deemed exclusionary by the investigator
11. Have had any other condition or are taking a medication that the investigator believes would interfere with the objectives of the study, pose a safety risk, or confound the interpretation of the study results.
12. Change in supplements, medication, or major diet in 30 days prior to enrolment and throughout the study.
13. Taking any supplements or vitamins notably known to affect cognitive function (e.g. Living Nutrition Cognitive, Viridian Cognitive Complex, ginkgo biloba, fish oil etc., list not exhaustive), or any psychotropic medications and products which interact with acetylcholine esterase and/or NMDA receptors (6-week washout before screening). Vitamin D and Calcium supplements permitted if on a stable dose for the previous 3 months.
14. Users of inhaled nicotine products such as cigarettes or vape products with an inconsistent recent history of consumption i.e., those who have taken up smoking/vaping in the 12 months prior to screening, or those who have either given up or re-started smoking or vaping in the 12 months prior to screening, or those who intend to significantly modify their use of inhaled nicotine products during their participation in the study.
15. Has received treatment involving experimental drugs in the past 3 months.
16. Have a malignant disease or any concomitant end-stage organ disease, which, in the Investigator's judgment, contraindicates participation in the study.
17. Individuals who, in the opinion of the investigator, are considered to be poor clinical attendees or unlikely for any reason to be able to comply with the trial.
18. Any Participant who is an employee of the study site or an Atlantia Clinical Trials employee or their close family member or a member of their household.

Ages: 55 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-09-18 (Estimated)

PRIMARY OUTCOMES:
Absolute change in Executive Function Score in the Mitocholine group compared to the Placebo group. | Baseline to end of intervention (week 16)
  Assessed by the verbal fluency, colour-word interference and trail making tests in the Delis-Kaplan Executive Function System
Absolute change in Homocysteine levels in the Mitocholine group compared to the Placebo group. | Baseline to end of intervention (week 16)
  Assessed by serum Homocysteine levels (umol/L)

SECONDARY OUTCOMES:
Change in Choline levels in the Mitocholine group compared to the Placebo group | Baseline to end of intervention (week 16)
  Assessed by Choline in blood
Change in S-adenosylmethionone (SAM) levels in the Mitocholine group compared to the Placebo group | Baseline to end of intervention (week 16)
  Assessed by S-adenosylmethionone (SAM) in blood
Change in Betaine levels in the Mitocholine group compared to the Placebo group | Baseline to end of intervention (week 16)
  Assessed by Betine in blood
Change in Memory outcomes (visual memory) in the Mitocholine group compared to the Placebo group | Baseline to end of intervention (week 16)
  Assessed by a Paired Associated Learning Task
Change in Memory outcomes (episodic memory) in the Mitocholine group compared to the Placebo group | Baseline to end of intervention (week 16)
  Assessed by a Word Recall Task
Change in Language outcomes in the Mitocholine group compared to the Placebo group | Baseline to end of intervention (week 16)
  Assessed by the Boston Naming Test

CONTACTS AND LOCATIONS:
Overall Officials: Steve Morrison, Study Director — Mitocholine Ltd
Locations (1):
- Atlantia Clinical Trials, Cork, Munster, Ireland

IPD SHARING:
Plan to Share IPD: No